CLINICAL TRIAL: NCT01763619
Title: Freedom® Cervical Disc Use In The Treatment of Cervical Degenerative Disc Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: AxioMed Spine Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR-300
Record Dates: First submitted 2013-01-04; First posted 2013-01-09 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Symptomatic Cervical Degenerative Disc Disease (DDD) From C3-C7
Keywords: Cervical DDD; DDD; degenerative disc disease; C3-C7
MeSH Terms: conditions — Dowling-Degos Disease; Intervertebral Disc Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Freedom Cervical Disc (Experimental)
  Interventions: Device: Freedom Cervical Disc

INTERVENTIONS:
Device: Freedom Cervical Disc

SUMMARY:
This study will collect clinical and radiographic data on the Freedom Cervical Disc to monitor the device's safety and performance as part of a post-market evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature males or females, aged 21 to 65 years old, inclusive.
* Single, or adjacent, 2-level degenerative disc disease at C3-C7, inclusive.
* Subject is a surgical candidate for an anterior approach to the cervical spine.
* Minimum of 6 weeks of unsuccessful conservative treatment.
* Subject with at least moderate preoperative pain and functional impairment
* Subject is mentally and physically able to comply with protocol, postoperative compliance instructions, and follow-up schedule through 2-years.
* Subject must understand and sign the written Informed Consent form.

Exclusion Criteria:

* Subject with axial neck pain only who does not demonstrate concurrent arm pain or progressive neurological deterioration (specifically numbness or muscle weakness in the arm).
* An active infection at the operative site or active systemic infection at the time of surgery.
* Known or suspected allergy to titanium, polyurethane, cobalt, chromium, molybdenum or silicone.
* Previous spinal fusion at the involved, or adjacent, cervical level(s).
* Congenital or acquired structural defect at the operative levels (s) or their immediately adjacent level(s).
* Significant osteoporosis in the cervical spine.
* The investigator should assess if the subject has any of the following conditions at the index or adjacent level(s) which excludes the subject from study participation:
* Cervical facet degeneration of the involved C3-C7 levels.
* Previous trauma to, or fusion in, the C3-C7 levels.
* Cervical instability at the index level(s) on neutral lateral or flexion/extension x-rays.
* Radiographic findings of a fused or total collapsed disc.
* Significant global cervical kyphosis (≥15º on Cobb angle measurement) or significant reversal of lordosis.
* Female of childbearing potential, pregnant, breast feeding, or interested in becoming pregnant in the next two years

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-02; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Safety of FCD | 6 months
  Monitor the safety (operative and post-operative adverse events through 6-months) of the FCD.
Performance of FCD | 6 months
  Monitor the performance (radiographic evaluation of segmental non-fusion and device function) of the FCD through 6-months post-operative period.

SECONDARY OUTCOMES:
Incidence of AEs | 2 year
  Examine the incidence of adverse events including device revision, removal or supplemental fixation through the 2-years post-operative period.
Neck/Arm Pain | 2 years
  Examine changes in neck and arm pain throughout the 2-years post-operative period.
Neurological function | 2 years
  Examine changes in subject neurological function throughout the 2-years post-operative period.
Subject Function | 2 years
  Examine changes in subject function throughout the 2-years post-operative period.
Radiographic Measurements | 2 years
  Examine changes in radiographic measurements of the target, adjacent and cervical segment levels from discharge through the 2-years.
Examine AEs | 2 years
  Examine all adverse events throughout the 2-years post-operative period

CONTACTS AND LOCATIONS:
Locations (5):
- Germany (3):
  - Universitatsklinikum Bonn, Bonn
  - Stadtisches Klinikum Gorlitz, Görlitz
  - Stadtisches Klinikum Karlsruhe, Karlsruhe
- Switzerland (2):
  - Klinik St. Anna, Lucerne
  - Spine Center Rischke, Zurich